CLINICAL TRIAL: NCT01008618
Title: A Verification Study of JNS020QD in Patients With Osteoarthritis or Low Back Pain
Brief Title: A Confirmatory Study of Fentanyl in Participants With Osteoarthritis or Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR015541; JNS020QD-JPN-N01
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Results first posted 2013-07-10 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Pain; Osteoarthritis; Low Back Pain
Keywords: Chronic pain; Osteoarthritis; Low back pain; Fentanyl; JNS020QD; Patch, transdermal; Opioid analgesics
MeSH Terms: conditions — Chronic Pain; Osteoarthritis; Low Back Pain | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fentanyl (Titration period) (Experimental): One-day adhesive transdermal patch containing fentanyl (JNS020QD) applied to chest, abdomen, upper arm and thigh and replaced every day, starting at the dose of 12.5 microgram per hour (mcg/hr) for at least first 2 days, which will be increased by 12.5 mcg/hr at one time based on the medical examination of number of rescue treatments and visual analog scale (VAS) score of the participants. The dose will be increased up to maximum of 50 mcg/hr. The treatment will be continued for 10-29 days and then the eligible participants from this group will be randomly assigned to either of the two groups in the double-blind period.
  Interventions: Drug: Fentanyl
- Fentanyl (Double-blind period) (Experimental): Participants meeting the pre-defined criteria for transfer from titration period to double-blind period and randomly assigned to fentanyl group, will be administered one-day adhesive transdermal patch containing fentanyl, applied to chest, abdomen, upper arm and thigh and replaced every day, the dose of which will be same as the final application dose in the titration period (in the range of 12.5 to 50 mcg/hr). The treatment will be continued for 12 weeks.
  Interventions: Drug: Fentanyl
- Placebo (Double-blind period) (Placebo Comparator): Participants meeting the pre-defined criteria for transfer from titration period to double-blind period and randomly assigned to placebo group, will be administered one-day adhesive transdermal placebo patch indistinguishable from fentanyl in appearance, applied to chest, abdomen, upper arm and thigh and replaced every day. The dose of fentanyl (from titration period) will be gradually decreased to prevent withdrawal symptoms and the dose of the matching placebo will be gradually increased up to same dose as the final application dose in the titration period (in the range of 12.5 to 50 mcg/hr). The treatment will continue for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fentanyl — One-day adhesive transdermal patch containing fentanyl 12.5 to 50 mcg/hr applied to chest, abdomen, upper arm or thigh and replaced every day.
  Arms: Fentanyl (Double-blind period); Fentanyl (Titration period)
Drug: Placebo — Placebo patch indistinguishable from one-day adhesive transdermal patch containing fentanyl 12.5 to 50 mcg/hr applied to chest, abdomen, upper arm or thigh and replaced every day.
  Arms: Placebo (Double-blind period)

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of fentanyl in opioid-naive participants with osteoarthritis (disorder, which is seen mostly in older persons, in which the joints become painful and stuff) or low back pain who cannot obtain a sufficient analgesic effect by the treatment of non-opioid analgesics (drug used to control pain).

DETAILED DESCRIPTION:
This is a multi-center (conducted in more than one center), double-blind (neither the participant nor the physician knows the assigned study drug), randomized (participants assigned study drug by chance), withdrawal study in opioid-naive participants with osteoarthritis or low back pain. The study will consist of titration period (10-29 days) and double-blind period (12 weeks) and the visits will include Day 5-7, 8, 15, 29 in titration period and Day 2-4, 8, 15, 22, 29, 43, 57, 71 and 85 in double-blind period. All the eligible participants will receive one-day adhesive transdermal patch (patch containing a drug that is put on the skin so the drug will enter the body through the skin) of either fentanyl at the dose ranging from 12.5 to 50 microgram per hour (mcg/hr) or matching placebo. Efficacy will be evaluated primarily by time to withdrawal due to insufficient analgesic efficacy. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants whose pain because of osteoarthritis or low back pain is continuing for at least 12 weeks prior to informed consent
* Participants who are continuously taking a non-opioid analgesic at the normal highest dose or more for at least 14 consecutive days prior to informed consent, or participant at a certain dose (except the use on an as-needed base) on consecutive days
* Participants showing insufficient therapeutic efficacy of the non-opioid analgesic currently being used, and requiring a continuous opioid analgesic as per the investigator or sub-investigator
* Participants with an average pain intensity of 50 millimeter or more on the Visual Analog Scale (VAS) in 24-hour daily living prior to informed consent
* Participants who can be hospitalized to the 4th day after the initiation of titration period

Exclusion Criteria:

* In cases of low back pain, participants with severe pain of lower extremities due to radiculopathy (a problem in which one or more nerves are affected) than that of low back pain, or participants with disc herniation (a medical condition affecting the spine due to trauma, lifting injuries, or idiopathic [unknown] causes) requiring an operation
* In cases of low back pain, participants with pain due to compression fracture
* Participants who had an operation that may affect the assessment within 30 days before informed consent
* Participants whose main cause of the pain to be assessed is considered attributable to psychogenic pain (physical pain that is caused, increased, or prolonged by mental, emotional, or behavioral factors)
* Participants with asthma, bradyarrhythmia (slow irregular heart beat) and severe respiratory function disorders

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2009-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (59):
- Japan (59):
  - Aki
  - Akō
  - Amagasaki
  - Anan
  - Annaka
  - Chiba
  - Chiisagata
  - Fuchū
  - Fukuoka
  - Fukuyama
  - Hamamatsu
  - Hiki
  - Himeji
  - Hiratsuka
  - Hitachi-Naka
  - Ichikawa
  - Ikeda
  - Ikoma
  - Itō
  - Izumo
  - Kagoshima
  - Kanazawa
  - Kasama
  - Kitakyushu
  - Kochi
  - Koga
  - Komatsu
  - Kure
  - Kurume
  - Kyoto
  - Maebaru
  - Matsudo
  - Matsumoto
  - Miyazaki
  - Nagano
  - Nagoya
  - Niihama
  - Ohkawa
  - Ohmuta
  - Ohta-Ku
  - Ohtsu
  - Osaka
  - Otaru
  - Ōita
  - Saga
  - Sagamihara
  - Sapporo
  - Sendai
  - Suginami-Ku
  - Takaoka
  - Takasaki
  - Takayama
  - Tatebayashi
  - Tokushima
  - Tokyo
  - Toshima-Ku
  - Toyama
  - Ube
  - Yokohama

REFERENCES:
- [Derived] Arai T, Kashimoto Y, Ukyo Y, Tominaga Y, Imanaka K. Two placebo-controlled, randomized withdrawal studies to evaluate the fentanyl 1 day patch in opioid-naive patients with chronic pain. Curr Med Res Opin. 2015 Dec;31(12):2207-18. doi: 10.1185/03007995.2015.1092127. Epub 2015 Oct 19. PMID 26359327

RESULTS

PARTICIPANT FLOW:
Groups:
- Fentanyl (Titration Period): One-day adhesive transdermal patch (patch containing a drug that is put on the skin so the drug will enter the body through the skin) containing fentanyl (JNS020QD) applied to chest, abdomen, upper arm or thigh and replaced every day, starting at the dose of 12.5 microgram per hour (mcg/hr) for at least first 2 days, which was increased by 12.5 mcg/hr at one time based on the medical examination of number of rescue treatments and visual analog scale (VAS) of the participants. The dose was increased up to maximum of 50 mcg/hr. The treatment was continued for 10-29 days and then the eligible participants from this group were randomly assigned to either of the two groups in the double-blind period.
- Fentanyl (Double-blind Period): Participants meeting the pre-defined criteria for transfer from titration period to double-blind period and randomly assigned to fentanyl group, were administered one-day adhesive transdermal patch containing fentanyl, applied to chest, abdomen, upper arm or thigh and replaced every day, the dose of which was same as the final application dose in the titration period (in the range of 12.5 to 50 mcg/hr). The treatment was continued for 12 weeks.
- Placebo (Double-blind Period): Participants meeting the pre-defined criteria for transfer from titration period to double-blind period and randomly assigned to placebo group, were administered one-day adhesive transdermal placebo patch indistinguishable from fentanyl in appearance, applied to chest, abdomen, upper arm or thigh and replaced every day. The dose of fentanyl (from titration period) was gradually decreased to prevent withdrawal symptoms and the dose of the matching placebo was gradually increased up to same dose as the final application dose in the titration period (in the range of 12.5 to 50 mcg/hr). The treatment was continued for 12 weeks.
Period: Period 1 (Titration Period)
Arm/Group | Fentanyl (Titration Period) | Fentanyl (Double-blind Period) | Placebo (Double-blind Period)
Started | 218 | 0 | 0
Completed | 150 | 0 | 0
Not Completed | 68 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Adverse Event | 33 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 0 | 0
Not completed — Not satisfied criteria to enter Period 2 | 20 | 0 | 0
Not completed — Aggravated symptom | 2 | 0 | 0
Period: Period 2 (Double-Blind Period)
Arm/Group | Fentanyl (Titration Period) | Fentanyl (Double-blind Period) | Placebo (Double-blind Period)
Started | 0 | 73 | 77
Completed | 0 | 37 | 39
Not Completed | 0 | 36 | 38
Not completed — Adverse Event | 0 | 11 | 2
Not completed — Withdrawal by Subject | 0 | 3 | 2
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Insufficient analgesic efficacy | 0 | 0 | 3
Not completed — More than 3 times a day rescue treatment | 0 | 0 | 1
Not completed — More than 15mm increase in Mean VAS | 0 | 21 | 29
Not completed — Not appropriate for this study | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Arm/Group | Fentanyl (Titration Period)
Number analyzed (Participants) | 218
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.8 (13.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145
  Male | 73

OUTCOME MEASURES:

1. Primary Outcome: Time From the Initial Day of Application in Double-Blind Period to Withdrawal Because of Insufficient Analgesic Efficacy
Description: Time from start of double-blind (researchers and participants were unaware of the treatment) period to withdrawal because of insufficient analgesic efficacy based on any of the pre-defined discontinuation criteria was noted.
Time Frame: Day 1 up to Day 85 (double-blind period) and Day 92 (discontinuation of the study)
Population: Full analysis set (FAS) population included all the randomly assigned participants with the exception of participants with pre-defined criteria.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Fentanyl (Double-blind Period): Participants meeting the pre-defined criteria for transfer from titration period to double-blind period and randomly assigned to fentanyl group, were administered one-day adhesive transdermal patch containing fentanyl, applied to chest, abdomen, upper arm and thigh and replaced every day, the dose of which was same as the final application dose in the titration period (in the range of 12.5 to 50 mcg/hr). The treatment was continued for 12 weeks.
- Placebo (Double-blind Period): Participants meeting the pre-defined criteria for transfer from titration period to double-blind period and randomly assigned to placebo group, were administered one-day adhesive transdermal placebo patch indistinguishable from fentanyl in appearance, applied to chest, abdomen, upper arm and thigh and replaced every day. The dose of fentanyl (from titration period) was gradually decreased to prevent withdrawal symptoms and the dose of the matching placebo was gradually increased up to same dose as the final application dose in the titration period (in the range of 12.5 to 50 mcg/hr). The treatment was continued for 12 weeks.
Arm/Group | Fentanyl (Double-blind Period) | Placebo (Double-blind Period)
Number analyzed (Participants) | 73 | 77
Days | NA [NA to NA] — The data was not estimable due to the high number of participants censored for this outcome measure. | NA [21.0 to NA] — The data was not estimable due to the high number of participants censored for this outcome measure.
Statistical Analysis 1: Comparison: Fentanyl (Double-blind Period) vs Placebo (Double-blind Period); Test type: Superiority or Other; p = 0.0846, Log Rank

2. Secondary Outcome: Pain Visual Analog Scale (VAS) Score - Titration Period
Description: The intensity of average pain (degree of pain) felt by the participants in daily living throughout the day on a "100-millimeter (mm) VAS scale" by drawing a slash. The left margin (0 mm) was considered "No pain at all", and the right margin (100 mm) was considered "Severer pain than this is inconceivable". The length (mm) from the left margin to the slash is measured. Mean VAS score during 3 days before the end of Screening period and during 3 days before the end of titration period was reported.
Time Frame: Day 12-14 (Screening period) and Day 27-29 (Titration period)
Population: Full analysis set in Period 1 (FAS1) population included all the randomly assigned participants with the exception of participants with pre-defined criteria. 'N' (number of participants analyzed) = participants evaluable for this measure and 'n' = participants evaluable for this measure at given time points.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Fentanyl (Titration Period): One-day adhesive transdermal patch (patch containing a drug that is put on the skin so the drug will enter the body through the skin) containing fentanyl (JNS020QD) applied to chest, abdomen, upper arm and thigh and replaced every day, starting at the dose of 12.5 microgram per hour (mcg/hr) for at least first 2 days, which was increased by 12.5 mcg/hr at one time based on the medical examination of number of rescue treatments and visual analog scale (VAS) score of the participants. The dose was increased up to maximum of 50 mcg/hr. The treatment was continued for 10-29 days and then the eligible participants from this group were randomly assigned to either of the two groups in the double-blind period.
Arm/Group | Fentanyl (Titration Period)
Number analyzed (Participants) | 218
mm
  Last 3 days in Screening period (n=218) | 74.1 (12.37)
  Last 3 days in titration period (n=216) | 39.71 (21.41)

3. Secondary Outcome: Pain Visual Analog Scale (VAS) Score - Double-Blind Period
Description: The intensity of average pain (degree of pain) felt by the participants in daily living throughout the day on a "100-millimeter (mm) VAS scale" by drawing a slash. The left margin (0 mm) was considered "No pain at all", and the right margin (100 mm) was considered "Severer pain than this is inconceivable". The length (mm) from the left margin to the slash is measured. Mean VAS score during 3 days before the end of titration period and during 3 days before the end of double-blind period was reported.
Time Frame: Day 27-29 (Titration period) and Day 83-85 (double-blind period)
Population: The FAS population included all the randomly assigned participants with the exception of participants with pre-defined criteria. 'N' (number of participants analyzed) = participants evaluable for this measure and 'n' = participants evaluable for this measure at given time points.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Fentanyl (Double-blind Period) | Placebo (Double-blind Period)
Number analyzed (Participants) | 73 | 77
mm
  Last 3 days in titration period (n=73, 77) | 28.9 (12.71) | 29.6 (12.05)
  Last 3 days in double-blind period (n=72, 77) | 28.9 (18.99) | 36.5 (22.29)

4. Secondary Outcome: Number of Participants Evaluated as Per Participant's Overall Assessment - Titration Period
Description: The participant assessed his/her satisfaction with the therapeutic efficacy by the following 5 grades: "Extremely satisfied", "Satisfied", "Neither satisfied nor dissatisfied", "Dissatisfied" and "Dissatisfied very much". The results were reported as Category 1 = At least "Neither satisfied nor dissatisfied", which included participants with general evaluation of "Extremely satisfied" to "Neither satisfied nor dissatisfied", and Category 2 = At least "Satisfied", which included participants with general evaluation of "Extremely satisfied" to "Satisfied".
Time Frame: Day 1 and 29 or final evaluation (Titration period)
Population: The FAS1 population included all the randomly assigned participants with the exception of participants with pre-defined criteria. 'N' (number of participants analyzed) = participants evaluable for this measure and 'n' = participants evaluable for this measure at given time points.
Measure: Number; unit: Participants
Groups:
- Fentanyl (Titration Period): One-day adhesive transdermal patch containing fentanyl applied to chest, abdomen, upper arm and thigh and replaced every day, starting at the dose of 12.5 mcg/hr for at least first 2 days, which was increased by 12.5 mcg/hr at one time based on the medical examination of number of rescue treatments and VAS score of the participants. The dose was increased up to maximum of 50 mcg/hr. The treatment was continued for 10-29 days and then the eligible participants from this group were randomly assigned to either of the two groups in the double-blind period.
Arm/Group | Fentanyl (Titration Period)
Number analyzed (Participants) | 218
Participants
  Day 1, Category 1 (n=218) | 77
  Day 1, Category 2 (n=218) | 11
  Day 29/Final evaluation, Category 1 (n=218) | 183
  Day 29/ Final evaluation, Category 2 (n=218) | 124

5. Secondary Outcome: Number of Participants Evaluated as Per Participant's Overall Assessment - Double-Blind Period
Description: as for outcome 4
Time Frame: Day 1 and 85 or final evaluation (double-blind period)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Fentanyl (Double-blind Period) | Placebo (Double-blind Period)
Number analyzed (Participants) | 73 | 77
Participants
  Day 1, Category 1 (n=73, 77) | 71 | 76
  Day 1, Category 2 (n=73, 77) | 57 | 63
  Day 85/Final evaluation, Category 1 (n=73, 77) | 63 | 56
  Day 85/Final evaluation, Category 2 (n=73, 77) | 42 | 35

6. Secondary Outcome: Number of Doses of Rescue Treatment Per Day - Titration Period
Description: If a breakthrough pain occurred or the analgesic efficacy became insufficient, a fast-acting oral morphine was administered. At such instances, one-time dose of the rescue treatment was administered as per the pre-defined criteria. During hospitalization, Investigator, Sub-investigator or Study Collaborator recorded in the medical record and during the out-patient period, the participants were instructed to describe the name of rescue treatment, date and time of treatment, and one-time dose in the participant's diary. The mean number of treatments per day at each assessment time was reported.
Time Frame: Day 1 and 29 or final evaluation (Titration period)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Treatments per day
Arm/Group | Fentanyl (Titration Period)
Number analyzed (Participants) | 218
Treatments per day
  Day 1 (n=218) | 0.0 (0.19) [0 to 3]
  Day 29/Final evaluation (n=218) | 0.2 (0.45)

7. Secondary Outcome: Number of Doses of Rescue Treatment Per Day - Double-Blind Period
Description: as for outcome 6
Time Frame: Day 1 and 85 or final evaluation (double-blind period)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Treatments per day
Arm/Group | Fentanyl (Double-blind Period) | Placebo (Double-blind Period)
Number analyzed (Participants) | 73 | 77
Treatments per day
  Day 1 (n=73, 77) | 0.0 (0.16) [0 to 2] | 0.0 (0.11) [0 to 2]
  Day 85/Final evaluation (n=72, 77) | 0.2 (0.49) | 0.2 (0.42)

8. Secondary Outcome: Brief Pain Inventory Short Form (BPI-sf) Score - Titration Period
Description: The BPI-sf total score is an average of the pain interference score (mean value for the nine BPI-sf questions [questions inquiring about the extent of interference with activities by pain, where the extent is ranked from 0 (does not interfere) to 10 (completely interferes)]) and pain subscale score (mean value for the scores for BPI-sf questions 3, 4, 5 and 6 [questions inquiring about the extent of pain, where the extent is ranked from 0 (no pain) to 10 (pain as bad as you can imagine)]). Total score ranges from 0 to 10 with higher values indicating more pain.
Time Frame: Day 1 and 29 or final evaluation (Titration period)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fentanyl (Titration Period)
Number analyzed (Participants) | 218
Units on a scale
  Day 1 (n=218) | 5.9 (1.66)
  Day 29/Final evaluation (n=217) | 4.0 (2.19)

9. Secondary Outcome: Brief Pain Inventory Short Form (BPI-sf) Score - Double-Blind Period
Description: as for outcome 8
Time Frame: Day 1 and 85 or final evaluation (double-blind period)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fentanyl (Double-blind Period) | Placebo (Double-blind Period)
Number analyzed (Participants) | 73 | 77
Units on a scale
  Day 1 (n=73, 77) | 3.2 (1.65) | 3.2 (1.66)
  Day 85/Final evaluation (n=73, 77) | 3.2 (1.83) | 3.9 (2.08)

10. Secondary Outcome: Short-Form 36-Item Health Survey Version 2.0 (SF-36v2) - Titration Period
Description: The SF-36v2 is 36-item form related to 8 health concepts (physical functioning, role physical, role emotional, general health, social functioning, bodily pain, vitality, mental health) and 2 summary scores (physical and mental component summary). Physical functioning, role physical and bodily pain contribute to physical component; role emotional, social functioning and mental health contribute to mental component; and social functioning, vitality, and general health contribute to both. All scores are based on a scale from 0 to 100, with higher scores defining more favorable health state.
Time Frame: Day 1 and 29 or final evaluation (Titration period)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fentanyl (Titration Period)
Number analyzed (Participants) | 218
Units on a scale
  Day 1, Physical Component Score (n=218) | 17.1 (14.91)
  Day 1, Mental Component Score (n=218) | 48.2 (9.92)
  Day 29/Final, Physical Component Score (n=217) | 23.3 (15.56)
  Day 29/Final, Mental Component Score (n=217) | 48.5 (9.57)

11. Secondary Outcome: Short-Form 36-Item Health Survey Version 2.0 (SF-36v2) - Double-Blind Period:
Description: as for outcome 10
Time Frame: Day 1 and 85 or final evaluation (double-blind period)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fentanyl (Double-blind Period) | Placebo (Double-blind Period)
Number analyzed (Participants) | 73 | 77
Units on a scale
  Day 1, Physical Component Score (n=73, 77) | 25.8 (14.71) | 22.8 (14.30)
  Day 1, Mental Component Score (n=73, 77) | 50.1 (8.29) | 50.8 (9.13)
  Day 85/Final, Physical Component Score (n=73, 77) | 24.3 (16.11) | 22.5 (14.64)
  Day 85/Final, Mental Component Score (n=73, 77) | 49.9 (9.82) | 51.0 (10.41)

12. Secondary Outcome: Number of Participants Evaluated as Per Physician's Overall Assessment - Titration Period
Description: Physician's global assessment of therapeutic efficacy (effectiveness) of the study drug was measured on a 2-point scale where 1 = effective and 2 = not effective.
Time Frame: Day 29 or final evaluation (Titration period)
Population: The FAS1 population included all the randomly assigned participants with the exception of participants with pre-defined criteria.
Measure: Number; unit: Participants
Arm/Group | Fentanyl (Titration Period)
Number analyzed (Participants) | 218
Participants
  Effective | 185
  Ineffective | 33

13. Secondary Outcome: Number of Participants Evaluated as Per Physician's Overall Assessment - Double-Blind Period
Description: as for outcome 12
Time Frame: Day 1 and 85 or final evaluation (double-blind period)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Fentanyl (Double-blind Period) | Placebo (Double-blind Period)
Number analyzed (Participants) | 73 | 77
Participants
  Day 1, Effective (n= 73, 77) | 73 | 77
  Day 1, Ineffective (n= 73, 77) | 0 | 0
  Day 85/Final evaluation, Effective (n= 73, 77) | 64 | 51
  Day 85/Final evaluation, Ineffective (n= 73, 77) | 9 | 26

ADVERSE EVENTS:
Time Frame: From Screening period up to the Follow-up period
Arm/Group | Fentanyl (Titration Period) | Fentanyl (Double-blind Period) | Placebo (Double-blind Period)
Serious Adverse Events (participants affected / at risk) | 12/218 | 3/73 | 2/77
Other Adverse Events (participants affected / at risk) | 177/218 | 50/73 | 35/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fentanyl (Titration Period) (N=218) | Fentanyl (Double-blind Period) (N=73) | Placebo (Double-blind Period) (N=77)
Nausea (Gastrointestinal disorders) | 3 | 0 | 0
Pain (General disorders) | 1 | 1 | 0
Positional vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Hallucinations (Psychiatric disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Chronic heart failure (Vascular disorders) | 1 | 0 | 0
Gastric discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Aspiration pneumonia (Infections and infestations) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Lassitude (General disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Death (General disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fentanyl (Titration Period) (N=218) | Fentanyl (Double-blind Period) (N=73) | Placebo (Double-blind Period) (N=77)
Nasopharyngitis (Infections and infestations) | 6 | 10 | 8
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0
Impetigo (Infections and infestations) | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis bacterial (Infections and infestations) | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2 | 5
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 5 | 7 | 3
Hallucination (Psychiatric disorders) | 3 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 1 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 59 | 3 | 0
Dizziness (Nervous system disorders) | 27 | 1 | 2
Headache (Nervous system disorders) | 15 | 0 | 1
Dysgeusia (Nervous system disorders) | 2 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0
Head discomfort (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 1
Myelopathy (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 0
Palpitations (Cardiac disorders) | 2 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Raynaud's phenomenon (Vascular disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 91 | 5 | 6
Constipation (Gastrointestinal disorders) | 66 | 6 | 3
Vomiting (Gastrointestinal disorders) | 29 | 3 | 1
Abdominal discomfort (Gastrointestinal disorders) | 11 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 9 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1
Eructation (Gastrointestinal disorders) | 1 | 0 | 0
Faeces hard (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 2 | 0
Periodontitis (Gastrointestinal disorders) | 1 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 4 | 0 | 2
Liver disorder (Hepatobiliary disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 0 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 6 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Xeroderma (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Dysuria (Renal and urinary disorders) | 2 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 0
Sexual dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0
Genital haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Application site pruritus (General disorders) | 12 | 0 | 0
Malaise (General disorders) | 9 | 3 | 3
Thirst (General disorders) | 4 | 0 | 3
Application site dermatitis (General disorders) | 3 | 1 | 1
Feeling abnormal (General disorders) | 3 | 1 | 1
Application site erythema (General disorders) | 2 | 1 | 0
Drug withdrawal syndrome (General disorders) | 2 | 4 | 1
Hypothermia (General disorders) | 2 | 0 | 0
Oedema (General disorders) | 2 | 0 | 0
Pyrexia (General disorders) | 2 | 2 | 1
Application site pain (General disorders) | 1 | 0 | 0
Application site rash (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 2 | 1
Temperature regulation disorder (General disorders) | 1 | 0 | 0
Sensation of foreign body (General disorders) | 1 | 0 | 0
Application site discomfort (General disorders) | 1 | 0 | 0
Blood pressure increased (Investigations) | 5 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 0 | 1
White blood cell count increased (Investigations) | 2 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 2
Blood pressure decreased (Investigations) | 1 | 0 | 0
Blood urea increased (Investigations) | 1 | 1 | 1
C-reactive protein increased (Investigations) | 1 | 0 | 0
Electrocardiogram ST segment elevation (Investigations) | 1 | 0 | 0
Glucose urine present (Investigations) | 1 | 1 | 0
Laboratory test abnormal (Investigations) | 1 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 2 | 1
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2
Extrapyramidal disorder (Nervous system disorders) | 0 | 1 | 0
Mental impairment (Nervous system disorders) | 0 | 0 | 1
Visual field defect (Nervous system disorders) | 0 | 0 | 1
Abnormal sensation in eye (Eye disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 1
Posterior capsule opacification (Eye disorders) | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 2 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis atrophic (Gastrointestinal disorders) | 0 | 1 | 0
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Piloerection (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Benign prostatic hyperplasia (Renal and urinary disorders) | 0 | 1 | 0
Application site reaction (General disorders) | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 1
Facial pain (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Injection site extravasation (General disorders) | 0 | 1 | 0
Irritability (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 0
Application site eczema (General disorders) | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 2
Blood potassium decreased (Investigations) | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0
Eosinophil count increased (Investigations) | 0 | 1 | 0
Blood urine present (Investigations) | 0 | 1 | 0
Monocyte count increased (Investigations) | 0 | 1 | 0
Protein urine present (Investigations) | 0 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other